CLINICAL TRIAL: NCT00413855
Title: Elective Laparoscopic Appendectomy for Chronic Right Lower Abdominal Pain; Outcome of a Prospective Randomized Double-Blind Controlled Surgical Trial
Brief Title: Laparoscopic Appendectomy for Chronic Right Lower Abdominal Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 9335
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-12

CONDITIONS: Chronic or Recurrent Appendicitis
Keywords: Abdominal pain; Appendectomy; Laparoscopy; Chronic appendicitis; Appendicopathy
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Appendicitis; Abdominal Pain | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2; Surgical Procedures, Operative

INTERVENTIONS:
Procedure: laparoscopic appendectomy or not (surgery)

SUMMARY:
It is questionable whether elective appendectomy can effectively reduce pain in persistent or recurrent lower abdominal quadrant pain due to chronic appendicitis.

A single centre randomised double-blind sham surgery controlled clinical trial studied the effects of elective laparoscopic appendectomy on postoperative pain perception in patients with persistent or recurrent lower abdominal quadrant pain on abdominal pain at 6 months postoperatively. Secondary outcome was the relation between clinical response and the appendix' histopathology. The analysis was performed on an intention-to-treat basis. Pain scores were compared using a Fisher's exact test.

DETAILED DESCRIPTION:
Forty patients were randomised, 18 patients had a laparoscopic appendectomy and 22 patients had a laparoscopic inspection only. The postoperative pain scores were significantly different favouring appendix removal (p < 0.01). Relative risk calculations indicated a 2.4 fold (95% CI: 1.3 - 4.0) greater chance of improving or becoming pain free after laparoscopic appendectomy. The number needed to treat was 2.2 patients (95% CI: 1.5 - 6.5). There was no significant relation between postoperative pain scores and histopathology findings.

Conclusions Chronic or recurrent appendicitis is a realistic clinical entity that can be treated successfully by elective appendectomy leading to significant pain reduction in properly selected cases. Histopathology of the removed appendix does not contribute to the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were between 15 and 45 years of age, and if they suffered from chronic or recurrent right lower abdominal quadrant pain for more than three months. They were to experience continuous pain, or should have endured at least one pain attack in the month prior to inclusion.

Exclusion Criteria:

* Exclusion criteria consisted of (a history of) chronic back pain, previous abdominal surgery (with the exception of diagnostic laparoscopies or a laparoscopic sterilization), specific gastro-intestinal entities (such as inflammatory bowel disease) and gynaecological disease (all female patients consulted a gynaecologist). Routine laboratory investigations included hemoglobin rate, serum leukocyte count and differentiation, C-Reactive Protein concentration, Erythrocyte Sedimentation Rate, faeces cultures and urine sedimentation. Barium contrast studies of the colon were done in all patients, abdominal ultrasound or enteroclysis on discretion. Finally, exclusion was possible when diagnostic laparoscopy revealed abnormalities (see below).

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 1994-09; Study Completion 2005-06

PRIMARY OUTCOMES:
Primary outcome: pain reduction
The primary outcome measure was pain scored by the blinded patient at 6 months postoperatively

SECONDARY OUTCOMES:
Secondary outcome: histopathology
The secondary outcome parameter was the relation between clinical improvement and histopathological findings of the removed appendices

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Roumen, PhD, MD, Principal Investigator — Maxima Medical Center

REFERENCES:
- [Background] de Kok HJ. Laparoscopic appendectomy: a new opportunity for curing appendicopathy. Surg Laparosc Endosc. 1992 Dec;2(4):297-302. PMID 1341549